CLINICAL TRIAL: NCT02103244
Title: Pharmacokinetics of Carboplatin After Adjusted Dosing for High BMI, Low Serum Creatinine, and Maximal Renal Function
Brief Title: Validation of an Adjusted Dosing Algorithm of Carboplatin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARBMI
Record Dates: First submitted 2014-03-26; First posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Cancer
Keywords: pharmacokinetics; safety
MeSH Terms: conditions — Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carboplatin (Experimental): An adjusted dosing algorithm will be applied to calculate the dose of carboplatin. in 24 patients blood will be obtained in order to determine the pharmacokinetics of carboplatin after adjusted dosing
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — carboplatin will be dosed according to newly developed dosing algorithm.

SUMMARY:
An adjusted dosing algorithm for the dosing of the anticancer drug carboplatin has been developed, that accounts for high BMI, low serum creatinine values and maximal calculated renal function. The hypothesis is that this new dosing algorithm provides a more accurate and safe dose than dosing according to the old standard of care.

DETAILED DESCRIPTION:
Carboplatin is an alkylating anticancer drug that is used for the treatment of various types of cancer, including non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), malignant mesothelioma, ovarian cancer, and breast cancer. It is mostly given in combination with other chemotherapeutic drugs, but it can also be given as single agent.

Since carboplatin is highly eliminated by the kidneys, the dose needs to be adjusted for renal dysfunction. Furthermore, as there is clear correlation between the area under the concentration-time curve (AUC) of carboplatin and haematological toxicity and response rate, carboplatin is dosed per target AUC. For this, the standard pharmacokinetic formula [dose = clearance carboplatin x target AUC] is used.

the clearance is typically calculated using the cockcroft and gault (C-G) formula. In patients with high weight, or very low serum creatinine values the C-G-formula may overestimate the renal function, resulting in a potential overdose of carboplatin. the new developed dosing algorithm to be studied adjusts for high BMI and low serum creatinine values, in order to provide a more safe dose of carboplatin

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven advanced NSCLC, SCLC or ovarian cancer
* to be treated with carboplatin with a target AUC of 4, 5 or 6
* age 18 years or older
* WHO performance status 0 - 2
* adequate bone marrow and liver function defined as

  * haemoglobin ≥ 6.0 mmol/L
  * white blood cell count ≥ 3.0 * 109/L
  * absolute neutrophil count (ANC) ≥ 1.5 * 109/L
  * platelets ≥ 100/L
  * bilirubin ≤ 1.5 times ULN
  * ALAT and ASAT ≤ 2.5 times ULN (in case of liver metastases ≤ 5.0 times ULN).
* estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Treatment with carboplatin with a target AUC of <4
* active clinically serious infection
* history of a kidney allograft
* pregnant
* patients not suitable for follow-up
* pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
to the determine the mean absolute precision error and the mean prediction error of the AUC of carboplatin after dosing carboplatin according to the new dosing algorithm | 1 year

SECONDARY OUTCOMES:
Assessment of the incidence and severity of all adverse events that occurred during treatment with carboplatin | 1 year
  Treatment with carboplatin is associated with adverse drug reactions. As an oncolytic drug, treatment with carboplatin may for example result in myelosupression, infections and/or gastro-intestinal toxicity, that may require hospitalization for treatment of toxicity.
  With the new dosing algorithm we hope to provide a better calculation of the appropriate dose for the individual patient, and thereby a safer treatment. Therefore, adverse events of treatment is an important secondary outcome measure that will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: P. MG Filius, PharmD PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands